CLINICAL TRIAL: NCT02509806
Title: Apatinib as Maintenance Therapy After First-line Chemotherapy(DC for 4 Cycles) in Postoperative Recurrence/Metastasis Progressive Gastric Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investgator, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G309
Record Dates: First submitted 2015-07-26; First posted 2015-07-28 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib Maintenance Therapy After First-line Chemotherapy (Experimental): Apatinib Mesylate Tablets 500 mg qd p.o. after DC First-line Chemotherapy (Docetaxel 60-85mg/m2 i.v. d1, Cisplatin 60-75mg/m2 i.v. d1, q21d）
  Interventions: Drug: Apatinib
- No Intervention After First-line Chemotherapy (No Intervention): No Intervention after DC First-line Chemotherapy (Docetaxel 60-85mg/m2 i.v. d1, Cisplatin 60-75mg/m2 i.v. d1, q21d）

INTERVENTIONS:
Drug: Apatinib — Apatinib Mesylate Tablets 500 mg qd p.o.
  Other Names: ATAN
  Arms: Apatinib Maintenance Therapy After First-line Chemotherapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of apatinib as maintenance therapy after first-line chemotherapy in Postoperative Recurrence / Metastasis Progressive Gastric Cancer.

DETAILED DESCRIPTION:
Eligible patients will receive apatinib treatment(500mg qd p.o. q28d) until until disease progression or intolerable toxicity or patients withdrawal of consent after 4 cycles of DC first-line chemotherapy or only DC first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to75 years old;
2. Histologically proven progressive gastric cancer. All pts were received D2 gastrectomy and recurrence / metastasis occured;
3. Complete 4 cycles DC first-line chemotherapy and no and no disease progression occurred. DC: Docetaxel 60-85mg/m2 iv d1, Cisplatin 60-75mg/m2 iv d1, q21d;
4. ECOG PS of 0-1;
5. Major organ function has to meet the following criteria:

   ANC ≥ 1.5 × 109 / L; HB ≥ 90g / L; PLT ≥ 100 × 109 / L; Bilirubin <1.5 times the upper limit of normal (ULN); ALT and AST <2.5 × ULN; liver metastases, if any, the ALT and AST<5 × ULN;
6. An expected survival of ≥ 3 months;
7. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug.
8. Patient has to voluntarily join the study and sign the Informed Consent Form for the study;

Exclusion Criteria:

1. Confirmed that apatinib and/or its accessories allergy;
2. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than ClassI; I-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class II cardiac dysfunction;
3. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
4. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;
5. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
6. Associated with CNS (central nervous system) metastases;
7. Pregnant or lactating women;
8. Pts with other malignant tumor within 5 years(except cured skin basal cell carcinoma and cervical carcinoma);
9. With psychotropic drug abuse history and can't get rid of or mental disorder patients;
10. Participated in other clinical trials within 4 weeks.
11. Pts received VEGFR inhibitor treatment(i.e. sorafenib, sunitinib);
12. Any other condition that might place the patient at undue risk or preclude a patient from completing the study;
13. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | An expected average of 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei, China